CLINICAL TRIAL: NCT05712876
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of CK-0045 Following Subcutaneous Administration in Healthy Participants and Otherwise Healthy Participants With Obesity
Brief Title: A Phase 1 Study to Investigate Safety, Tolerability, and Pharmacokinetics of CK-0045 in Healthy Participants and Otherwise Healthy Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytoki Pharma (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CK-0045_CS01; 2022-002994-27 (EudraCT Number)
Record Dates: First submitted 2023-01-16; First posted 2023-02-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: Interleukin-22; Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single ascending dose (SAD) CK-0045 Dose level 1 to 5 (Experimental): At each dose level 6 healthy participants will receive a single dose of CK-0045 by s.c. administration
  Interventions: Drug: CK-0045
- SAD placebo (Placebo Comparator): At each dose level 2 healthy participants will receive a single dose of matching placebo by s.c. administration
  Interventions: Drug: Placebo
- Multiple ascending dose (MAD) CK-0045 Dose level 1 to 3 (Experimental): At each dose level 9 otherwise healthy participants with obesity will receive a loading dose of CK-0045 on Day 1 followed by a dose on Day 8, Day 15, Day 22, Day 29 and Day 36 of CK-0045 by s.c. administration
  Interventions: Drug: CK-0045
- MAD placebo (Placebo Comparator): At each dose level 3 otherwise healthy participants with obesity will receive matching placebo on Day 1, Day 8 , Day 15, Day 22, Day 29 and Day 36 by s.c. administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CK-0045 — Interleukin-22 agonist
  Arms: Multiple ascending dose (MAD) CK-0045 Dose level 1 to 3; Single ascending dose (SAD) CK-0045 Dose level 1 to 5
Drug: Placebo — Matching placebo
  Arms: MAD placebo; SAD placebo

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability and blood levels following a single dose or after multiple doses of CK-0045 given subcutaneously to healthy participants or otherwise healthy participants with obesity. 76 participants will receive CK-0045 or matching placebo at different escalating doses in 2 study parts: 40 healthy participants will receive a single dose and 36 otherwise healthy participants with obesity will receive 6 doses one week apart.

ELIGIBILITY:
Inclusion Criteria:

* For non-vasectomized men with partners who are women of child bearing potential (WOCBP) and for WOCBP, highly effective contraception for 3 months.
* For all female participants: a negative serum (β-hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1.
* In the opinion of the investigator, healthy based on medical history, physical and neurological examination, vital signs, and ECG, and clinical chemistry, hematology, coagulation, and urinalysis.
* A body weight in the range of 50 to 100 kg and a body mass index (BMI) of 18.5 to 27.0 kg/m2, inclusive, at screening for the SAD part and a BMI of 30.0 to 39.9 kg/m2, inclusive, at screening for the MAD part.
* A systolic blood pressure of ≥91 and ≤140 mmHg (SAD) / ≤145 mmHg (MAD) , a diastolic blood pressure of ≥51 and ≤80 mmHg (SAD) / ≤90 mmHg (MAD), and a pulse rate of ≥45 and ≤100 bpm at screening and Day 1 predose.
* Negative COVID-19 test (PCR) and no clinical symptoms of corona on Day -1.
* Signed informed consent form.
* Willing to adhere to the prohibitions and restrictions specified in the protocol.

Exclusion Criteria:

* Currently have or have a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant.
* Have one or more clinical laboratory test values outside the normal range at screening or on Day -1 (exceptions apply to MAD for fasting glucose, triglycerides, total cholesterol and liver enzymes).
* Has a QTcF interval >430 ms at screening or Day 1 predose for the SAD part or has a QTcF interval >450 ms (for male participants) or >470 ms (for female participants) at screening or Day 1 predose for the MAD part.
* Have a clinically significant or chronic infection or diagnosed latent infection.
* Significant acute illness within 7 days prior to the (first) study drug administration or have had a major illness or hospitalization within 1 month prior to the (first) study drug administration.
* Any history of clinically relevant skin diseases including but not limited to: Psoriasis, vitiligo, atopic dermatitis, eczema.
* History of any malignancy.
* Tattoos present on place of injection site.
* Major or traumatic surgery within 6 months of screening.
* Any participant who plans to undergo elective surgery within 4 weeks prior to the (first) study drug administration and through the end of the study.
* Positive serology test for HIV type 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies at screening.
* Recent history (within 6 months from screening) of alcohol or drug abuse.
* Active smoker and/or has used nicotine or nicotine-containing products (including e cigarettes or the equivalent of e-cigarettes) within the past 6 months of the (first) study drug administration.
* A positive urine toxicology screen at screening or Day -1 for substances of abuse.
* Have a positive alcohol breath test at screening or Day -1.
* Consumes, on average, more than approximately 500 mg/day of caffeine at screening for the SAD part or consumes, on average, more than approximately 700 mg/day of caffeine at screening for the MAD part.
* Donated blood within 90 days prior to (first) study drug administration.
* Trains/exercises intensively, e.g., for a marathon or triathlon, or at a competitive level.
* Have a history of active drug and/or food allergy or other active allergic disease requiring the constant use of medications, or a history of severe allergic reaction, angioedema or anaphylaxis at screening.
* Received any experimental therapy or new investigational agent within 30 days or 5 half-lives (whichever is longer) of the (first) study drug administration.
* Treatment with over-the-counter medications, and herbal medication within 14 days or prescription medications within 14 days or 5 half-lives (whichever is longer) prior to (first) study drug administration and through the end of the study, unless approved by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and seriousness of treatment emergent adverse events | Up to 8 weeks after last dose
  The safety and tolerability following single and multiple ascending doses of CK-0045 will be assessed

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Day 1 to 8 weeks after last dose
  The Cmax following single and multiple ascending doses of CK-0045 will be characterized
Area under the serum concentration-time curve from 0 to 168 hours (AUC168) after administration | Day 1 to Day 8
  AUC168 following single and multiple ascending doses of CK-0045 will be characterized
Area under the serum concentration-time curve from 0 to infinity (AUCinf) | Day 1 to 8 weeks after last dose
  AUCinf following single and multiple ascending doses of CK-0045 will be characterized

CONTACTS AND LOCATIONS:
Overall Officials: Anne Louise Kjølbye, PhD, Study Director — Cytoki Pharma; Lotte Verwillingen, MD, Principal Investigator — SGS Clinical Research, Clinical Pharmacology Unit
Locations (1):
- SGS Clinical Research, Clinical Pharmacology Unit, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No